CLINICAL TRIAL: NCT04287127
Title: Cosmetic Satisfaction and Undercorrection After One-stage Bone Lengthening in the Management of Brachymetatarsia
Brief Title: One-stage Bone Lengthening in the Management of Brachymetatarsia
Acronym: BRACHYONESTAGE
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0037
Record Dates: First submitted 2020-02-05; First posted 2020-02-27 (Actual); Last update posted 2020-03-02 (Actual); Status verified 2020-02

CONDITIONS: Brachymetatarsia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Brachymetatarsia is a shortening in length of a metatarsal exceeding 5mm. This congenital anomaly most often affecting women and the second metatarsal is associated with frequent aesthetic disorders leading patients to consult. The one-time lengthening technique is described for the management of brachymetatarsia with good functional results. However, the metatarsal elongation in one time is limited to 15 millimeters, to avoid complications.

No study has presented the consequences of hypocorrection, especially cosmetic. Our hypothesis is that undercorrection (Hypocorrection) is associated with a higher rate of cosmetic dissatisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients operated on for a one-time lengthening for isolated brachymetatarsia
* Major patients

Exclusion Criteria:

* Patient refusing to participate in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who presented brachymetatarsia and who underwent one stage lengthening in our department
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
satisfaction using a visual analog scale (from 0/10 to 10/10) | 1 day
  Cosmetic evaluation

SECONDARY OUTCOMES:
radiological evaluation of surgical correction | 1 day
  metatarsal lengtening : mesured on a dorsoplantar radiograph

CONTACTS AND LOCATIONS:
Overall Officials: Louis Dagneaux, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC